CLINICAL TRIAL: NCT00543868
Title: MK0782 + Low-Dose Aspirin 7-Day Erosion Endoscopy Study (0782-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0782-001; 2007_637
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Stomach Ulcer; Duodenal Ulcer
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0782

SUMMARY:
This study will determine how if MK0782 is safe and tolerable and to determine how often and the severity of stomach and small intestine ulcers develop following administration of MK0782 plus enteric coated aspirin, rofecoxib 25mg plus enteric coated aspirin, naproxen 500 mg puls enteric coated asprin vs placebo.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female
* 18 years of age or older (age at consent)
* Able to abstain from alcohol, tobacco, spicy foods, limit coffee
* Able to avoid strenuous activity
* Able to read and fill out a study diary

Exclusion Criteria:

* You have participated in an investigational drug study within 4 weeks of entering this study
* Your weight is not within a specific range for the study
* You have a history of GI problems like a gastric ulcer
* You have had gastric or intestinal surgery
* You have had abdominal or chest surgery
* You are currently abusing drugs or alcohol or have a history of abuse
* You have a history of psychiatric disorders
* You are a smoker or have smoked during the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2004-06; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC